CLINICAL TRIAL: NCT00586924
Title: A Phase I, Multicenter, Dose Escalation Study of CAT-8015 in Patients With Relapsed or Refractory Hairy Cell Leukemia (HCL)
Brief Title: A Phase I, Multicenter Dose Escalation Study in Patients With Hairy Cell Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Cambridge Antibody Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAT-8015-1001
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2018-12

CONDITIONS: Hairy Cell Leukemia
Keywords: CAT-8015; Moxetumomab pasudotox
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — immunotoxin HA22

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 5 mcg/kg (Experimental): Participants received intravenous infusion of 5 microgram per kilogram (mcg/kg) moxetumomab pasudotox (CAT-8015) on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until complete response (CR), progressive disease (PD), initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Interventions: Drug: Moxetumomab Pasudotox (CAT 8015)
- 10 mcg/kg (Experimental): Participants received intravenous infusion of 10 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Interventions: Drug: Moxetumomab Pasudotox (CAT 8015)
- 20 mcg/kg (Experimental): Participants received intravenous infusion of 20 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Interventions: Drug: Moxetumomab Pasudotox (CAT 8015)
- 30 mcg/kg (Experimental): Participants received intravenous infusion of 30 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Interventions: Drug: Moxetumomab Pasudotox (CAT 8015)
- 40 mcg/kg (Experimental): Participants received intravenous infusion of 40 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Interventions: Drug: CAT 8015 (Moxetumomab Pasudotox)
- 50 mcg/kg (Experimental): Participants received intravenous infusion of 50 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Interventions: Drug: Moxetumomab Pasudotox (CAT 8015)

INTERVENTIONS:
Drug: Moxetumomab Pasudotox (CAT 8015) — Participants received intravenous infusion of 5 microgram per kilogram (mcg/kg) moxetumomab pasudotox (CAT-8015) on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until complete response (CR), progressive disease (PD), initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Arms: 5 mcg/kg
Drug: Moxetumomab Pasudotox (CAT 8015) — Participants received intravenous infusion of 10 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Arms: 10 mcg/kg
Drug: Moxetumomab Pasudotox (CAT 8015) — Participants received intravenous infusion of 20 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Arms: 20 mcg/kg
Drug: Moxetumomab Pasudotox (CAT 8015) — Participants received intravenous infusion of 30 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Arms: 30 mcg/kg
Drug: CAT 8015 (Moxetumomab Pasudotox) — Participants received intravenous infusion of 40 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Arms: 40 mcg/kg
Drug: Moxetumomab Pasudotox (CAT 8015) — Participants received intravenous infusion of 50 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
  Arms: 50 mcg/kg

SUMMARY:
A dose-escalation study to identify the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD), defined as the highest dose that can safely be given to a participant and establish the safest dose based on the highest tolerated dose for clinical testing.

DETAILED DESCRIPTION:
A Phase 1, multicenter, dose escalation study of moxetumomab pasudotox (CAT-8015) in participants with relapsed or refractory hairy cell leukemia (HCL) to estimate the MTD, defined as the highest dose that can be safely administered to a patient, and to establish a safe dose, based on the MTD, for subsequent clinical testing (Phase 2 recommended dose).

ELIGIBILITY:
Inclusion Criteria: Confirmed diagnosis of HCL, Measurable disease, Participant's must have had at least 2 prior systemic therapies. There must have been at least 2 prior courses of purine analog, or 1 if the response to this course lasted less than (<) 2 years, or if the participant had unacceptable toxicity to purine analog, Eastern Cooperative Oncology Group (ECOG) performance status of 0-2, Participant's with other cancers who meet eligibility criteria and have less than 5 years of disease free survival will be considered on a case-by-case basis, Life expectancy of greater than 6 months, as assessed by principal investigator, Must be able to understand and sign informed consent, Must be at least 18 years old, Female and male participants must agree to use an approved method of contraception during the study.

Exclusion Criteria: - History of allogeneic bone marrow transplant, Documented and ongoing central nervous system involvement with their malignant disease (history of central nervous system (CNS) involvement is not an exclusion criteria), Pregnant or breast-feeding females, HIV positive serology (due to increased risk of severe infection and unknown interaction of CAT-8015 with antiretroviral drugs, Hepatitis B surface antigen positive. - Hepatic function: Serum transaminases (either alanine transaminase (ALT) or aspartate transaminase (AST)) or bilirubin: greater than or equal to (>=) Grade 2, unless bilirubin is due to Gilbert's disease. -Renal function: Serum creatinine clearance less than or equal to (<=) 60 millilitre per minute (mL/min) as estimated by Cockroft-Gault formula. -Hematologic function: The absolute neutrophil count (ANC) < 1000/ cubic millimetres (cmm), or platelet count <50,000/cmm, if these cytopenias are not judged by the investigator to be due to underlying disease (i.e. potentially reversible with anti-neoplastic therapy). -Pulmonary function: Participant's with < 50% of predicted forced expiratory volume (FEV1) or <50% of predicted diffusing capacity for carbon monoxide (DLCO), corrected for hemoglobin concentration and alveolar volume. Uncontrolled pulmonary infection, presence of pulmonary edema, Oxygen saturation at rest < 88% measured by pulse oximetry or partial pressure of oxygen (PaO2) < 55 millimetre(s) of mercury (mm Hg), Serum albumin < 2 g/dL, Radioimmunotherapy within 2 years prior to enrollment in study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-05-10 (Actual); Primary Completion 2015-05-06 (Actual); Study Completion 2015-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (4):
- United States (3):
  - Research Site, Stanford, California
  - Research Site, Chicago, Illinois
  - Research Site, Bethesda, Maryland
- Research Site, Lodz, Poland

REFERENCES:
- [Result] Kreitman RJ, Tallman MS, Robak T, Coutre S, Wilson WH, Stetler-Stevenson M, Fitzgerald DJ, Lechleider R, Pastan I. Phase I trial of anti-CD22 recombinant immunotoxin moxetumomab pasudotox (CAT-8015 or HA22) in patients with hairy cell leukemia. J Clin Oncol. 2012 May 20;30(15):1822-8. doi: 10.1200/JCO.2011.38.1756. Epub 2012 Feb 21. PMID 22355053
- [Derived] Kreitman RJ, Tallman MS, Robak T, Coutre S, Wilson WH, Stetler-Stevenson M, FitzGerald DJ, Santiago L, Gao G, Lanasa MC, Pastan I. Minimal residual hairy cell leukemia eradication with moxetumomab pasudotox: phase 1 results and long-term follow-up. Blood. 2018 May 24;131(21):2331-2334. doi: 10.1182/blood-2017-09-803072. Epub 2018 Feb 27. PMID 29487070

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 mcg/kg: Participants received IV 5 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued until complete response (CR), progressive disease (PD), initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
- 10 mcg/kg: Participants received IV 10 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
- 20 mcg/kg: Participants received IV 20 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
- 30 mcg/kg: Participants received IV 30 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
- 40 mcg/kg: Participants received IV 40 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
- 50 mcg/kg: Participants received IV 50 mcg/kg moxetumomab pasudotox on Days 1, 3, and 5 of every 28-day cycle and continued cycles of therapy until CR, PD, initiation of alternative anticancer therapy, unacceptable toxicity, development of neutralizing antibodies, or another reason to discontinue therapy.
Period: Overall Study
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Started | 3 | 3 | 3 | 3 | 4 | 33
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 4 | 33
Not completed — Adverse event/serious adverse event | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Initiation of alternative cancer therapy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Disease progression | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Development of neutralizing antibodies | 2 | 2 | 2 | 0 | 0 | 22
Not completed — Complete response | 0 | 1 | 0 | 0 | 2 | 2
Not completed — Other | 1 | 0 | 1 | 1 | 1 | 6

BASELINE CHARACTERISTICS:
Population: Safety population: included all participants who received any treatment of moxetumomab pasudotox
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 56.3 (14.2) | 54.3 (6.1) | 56.3 (3.1) | 58.3 (4.0) | 61.8 (11.1) | 55.8 (9.0) | 56.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1 | 1 | 5 | 8
  Male | 2 | 3 | 3 | 2 | 3 | 28 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Adverse events are suspected of causal relationship to drug and are >=Grade (G) 3 in severity considered DLTs: G 3 or 4 hematologic abnormalities at baseline due to disease were not evaluable for hematologic DLT, G 2 allergic reactions of bronchospasm or urticaria, or any >= G3 allergic reaction, in presence of pre-medication were considered DLTs. Following >= G 3 non-hematological treatment-related toxicities not considered DLTs: Tumor lysis syndrome, G 3 low electrolyte levels with pre-existing low levels of same electrolytes, anticoagulant therapy, G 3 or 4 infection or neutropenic fever unless relationship to IP is suspected, G 3 transaminase, alkaline phosphatase, bilirubin or other liver function test elevation provided resolution to values required for study entry prior to start of next cycle, G 3 fever, G 3 hypertriglyceridemia and hypercholesterolemia, and G 4 hypertriglyceridemia lasting <2 months, G 3 hypoalbuminemia lasting <7 days occurred in absence of CLS.
Time Frame: Cycle 1 Day 1 to Cycle 2 Day 10 (each cycle duration was 28 days)
Population: Evaluable population for DLT included all participants who received any treatment of moxetumomab pasudotox, completed at least Cycle 2 Day 10, or discontinued treatment due to a DLT on or before Cycle 2 Day 10.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: The TEAEs are defined as adverse events (AEs) present at baseline that worsened in intensity after administration of investigational product or events absent at baseline that emerged after administration of study drug, for the period extending to 30 days after the last dose of study drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening situation (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received moxetumomab pasudotox.
Time Frame: From start of study drug administration until 30 days after the last dose of study drug (approximately 8 years)
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
Participants
  TEAEs | 3 | 3 | 3 | 3 | 4 | 33
  TESAEs | 0 | 0 | 0 | 2 | 0 | 4

3. Primary Outcome: Number of Participants With Vital Signs Abnormalities Recorded as Treatment-Emergent Adverse Events (TEAEs)
Description: Vital signs abnormalities reported as TEAEs included pyrexia, weight increased, dyspnoea, hypoxia, hypertension, hypotension.
Time Frame: From start of study drug administration until 30 days after the last dose of study drug (approximately 8 years)
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
Participants
  Pyrexia | 1 | 1 | 2 | 3 | 1 | 16
  Weight increased | 1 | 0 | 0 | 0 | 0 | 6
  Dyspnoea | 1 | 0 | 0 | 1 | 0 | 6
  Hypoxia | 0 | 0 | 0 | 1 | 0 | 1
  Hypertension | 0 | 1 | 0 | 1 | 0 | 0
  Hypotension | 0 | 0 | 0 | 2 | 0 | 10

4. Primary Outcome: Number of Participants With Clinically Relevant Electrocardiogram (ECG) Abnormalities Recorded as Adverse Events (AEs)
Description: Cardiac AEs observed in participants with clinically significant ECG abnormalities included; ECG QT prolonged, Sinus tachycardia and Atrioventricular block first degree.
Time Frame: From start of study drug administration until 30 days after the last dose of study drug (approximately 8 years)
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
Participants
  ECG QT prolonged | 1 | 0 | 0 | 2 | 0 | 2
  Sinus tachycardia | 0 | 0 | 0 | 1 | 0 | 2
  Atrioventricular block first degree | 0 | 0 | 0 | 0 | 1 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Recorded as Treatment-Emergent Adverse Events (TEAEs)
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as an adverse event.
Time Frame: From start of study drug administration until 30 days after the last dose of study drug (approximately 8 years)
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
Participants
  Alanine aminotransferase increased | 1 | 1 | 1 | 3 | 2 | 25
  Aspartate aminotransferase increased | 2 | 1 | 1 | 2 | 1 | 24
  Blood alkaline phosphatase increased | 0 | 0 | 0 | 1 | 0 | 5
  Blood bicarbonate decreased | 0 | 0 | 0 | 0 | 0 | 5
  Blood bilirubin increased | 2 | 1 | 1 | 0 | 1 | 2
  Blood creatine phosphokinase increased | 0 | 1 | 0 | 1 | 0 | 4
  Blood creatinine increased | 1 | 0 | 0 | 1 | 0 | 11
  Blood triglycerides increased | 0 | 1 | 0 | 1 | 1 | 2
  Gamma-glutamyltransferase increased | 0 | 0 | 0 | 1 | 0 | 7
  Blood uric acid increased | 1 | 0 | 0 | 1 | 0 | 1
  Hyperglycaemia | 2 | 0 | 0 | 2 | 2 | 13
  Hypermagnesaemia | 0 | 0 | 0 | 0 | 1 | 12
  Hypernatraemia | 0 | 0 | 0 | 0 | 0 | 6
  Hypertriglyceridaemia | 0 | 0 | 1 | 0 | 0 | 19
  Hyperuricaemia | 0 | 0 | 0 | 0 | 0 | 4
  Hypoalbuminaemia | 2 | 1 | 1 | 3 | 3 | 25
  Hypocalcaemia | 0 | 0 | 0 | 1 | 1 | 11
  Hypoglycaemia | 1 | 1 | 0 | 0 | 1 | 1
  Hypokalaemia | 0 | 0 | 0 | 2 | 0 | 2
  Hypomagnesaemia | 0 | 0 | 1 | 1 | 1 | 7
  Hyponatraemia | 0 | 0 | 0 | 2 | 3 | 7
  Hypophosphataemia | 0 | 0 | 0 | 1 | 0 | 10
  Hemoglobin urine | 0 | 0 | 0 | 1 | 0 | 0
  Protein urine | 0 | 0 | 0 | 0 | 1 | 1
  Proteinuria | 0 | 0 | 0 | 0 | 0 | 9
  Hemoglobinuria | 0 | 0 | 0 | 0 | 0 | 3
  Hypercholesterolaemia | 0 | 0 | 0 | 0 | 0 | 9
  Hyperkalaemia | 0 | 1 | 0 | 0 | 1 | 5
  Lymphopenia | 2 | 0 | 2 | 0 | 0 | 25
  White blood cell count decresed | 2 | 1 | 2 | 1 | 2 | 17
  Lymphocyte count decreased | 0 | 1 | 1 | 2 | 2 | 5
  Neutrophil count decreased | 2 | 0 | 0 | 0 | 0 | 10
  Hemoglobin decreased | 2 | 0 | 2 | 1 | 1 | 9
  Platelet count decreased | 1 | 0 | 0 | 0 | 2 | 6
  Haptoglobin decreased | 0 | 0 | 0 | 1 | 1 | 7

6. Primary Outcome: Number of Participants With Objective Response Rate (ORR): Complete Response (CR) or Partial Response (PR)
Description: Objective response rate defined as proportion of participants with confirmed CR or confirmed PR according to Response Evaluation Criteria for hairy cell leukemia (HCL). A CR is defined as: No evidence of leukemic cells by routine H/E stains of peripheral blood and bone marrow. No hepatomegaly, splenomegaly, or lymphadenopathy by physical examination and/or appropriate radiographic techniques. Normal complete blood count as: Neutrophils >= 1,500/mcL, Platelets >= 100,000/mcL, and Hemoglobin >= 11.0 gm/dL without transfusions or growth factors for at least 4 weeks. Partial response requires all of following: >=50% reduction in peripheral blood lymphocyte from pretreatment baseline value, lymphadenopathy, and abnormal hepatosplenomegaly by CT scan or physical exam, and complete blood count as Neutrophils >= 1,500/mcL, Platelets >=100,000/mcL, and Hemoglobin >= 11.0 g/dL or 50% improvement of all parameters over baseline without transfusions or growth factors for at least 4 weeks.
Time Frame: From Baseline (predose of Cycle 1 Day 1) through end of study (until CR, PD, initiation of alternative therapy, unacceptable toxicity, development of neutralizing antibodies, or other study discontinuation reasons) (approximately 8 years)
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
Participants | 3 | 3 | 2 | 2 | 3 | 29

7. Primary Outcome: Number of Participants With Complete Response (CR)
Description: The CR is defined by: No evidence of leukemic cells by routine H/E stains of the peripheral blood and bone marrow. No hepatomegaly, splenomegaly, or lymphadenopathy by physical examination and/or appropriate radiographic techniques. Normal complete blood count as exhibited by: Neutrophils >= 1,500/microliter (mcL), Platelets >= 100,000/mcL, and Hemoglobin >= 11.0 gram per deciliter (gm/dL) without transfusions or growth factors for at least 4 weeks.
Time Frame: as for outcome 6
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
Participants | 0 | 2 | 2 | 1 | 2 | 21

8. Primary Outcome: Number of Participants With Partial Response (PR)
Description: Partial response requires all of the following: >=50% decrease in peripheral blood lymphocyte count from the pretreatment baseline value, >=50% reduction in lymphadenopathy, >=50% reduction in abnormal hepatosplenomegaly by computed tomography or physical exam, Neutrophils >= 1,500/mcL or 50% improvement over baseline without growth factors for at least 4 weeks, Platelets >=100,000/mcL or 50% improvement over baseline, and Hemoglobin >= 11.0 g/dL or 50% improvement over baseline without transfusions or growth factors for at least 4 weeks. For participants who are transfusion-dependent at baseline, a hemoglobin of >= 9.0 g/dL without transfusions or growth factors for at least 4 weeks.
Time Frame: as for outcome 6
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
Participants | 3 | 1 | 0 | 1 | 1 | 8

9. Primary Outcome: Number of Participants With Stable Disease (SD)
Description: Stable disease was characterized by not meeting the criteria for CR, PR or PD.
Time Frame: as for outcome 6
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
Participants | 0 | 0 | 1 | 1 | 0 | 4

10. Primary Outcome: Number of Participants With Progressive Disease (PD)
Description: Progressive disease is defined by at least one of the following compared to pretreatment:>= 25% increase in the sum of the products of the greatest perpendicular dimensions of at least two lymph nodes on two consecutive examinations at least 2 weeks apart (at least 1 node must be >= 2 cm) or appearance of new palpable lymph nodes, >=25% increase in the size of the liver and/or spleen as determined by measurement below the respective costal margin, or appearance of new palpable hepatomegaly or splenomegaly that was not previously present, >=50% increase in the absolute number of circulating lymphocytes, >=25% decrease in hemoglobin (must be < 11g/dL), platelets (must be < 100,000/mcL), or absolute neutrophil count (must be < 1500/mcL) unless these are judged to be effects of treatment.
Time Frame: as for outcome 6
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
Participants | 0 | 0 | 0 | 0 | 1 | 0

11. Primary Outcome: Time to Complete Response
Description: Time to complete response (CR) was measured from the start of moxetumomab pasudotox treatment to the first documentation of CR and was evaluated only in participants who received any treatment of moxetumomab pasudotox and had achieved a CR. Time to complete response was summarized using Kaplan-Meier estimates (median time, 95% confidence interval [CI] for median time).
Time Frame: as for outcome 6
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox. The "Overall Number of Participants Analyzed" denotes the number of participants who had achieved a CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 0 | 2 | 2 | 1 | 2 | 21
months |  | 2.53 [2.30 to 2.76] | 9.56 [4.11 to 15.01] | 3.71 [3.71 to 3.71] | 2.53 [2.27 to 2.79] | 3.94 [2.30 to 6.31]

12. Primary Outcome: Time to Objective Response
Description: Time to OR was measured from the start of moxetumomab pasudotox treatment to the first documentation of OR and was evaluated only in participants who received any treatment of moxetumomab pasudotox and had achieved an OR (CR or PR). Objective response (OR) was defined as the participants with confirmed CR or confirmed PR according to Response Evaluation Criteria.
Time Frame: as for outcome 6
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox. The "Overall Number of Participants Analyzed" denotes the number of participants who had achieved an OR (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 2 | 2 | 3 | 29
months | 3.02 [2.04 to 4.80] | 1.12 [0.92 to 2.76] | 8.2 [1.38 to 15.01] | 8.18 [1.87 to 14.49] | 1.08 [0.95 to 2.79] | 1.05 [0.92 to 1.58]

13. Primary Outcome: Duration of Complete Response
Description: Duration of CR was measured from the first documentation of CR to the first documented non-CR and was evaluated in participants who had achieved an CR. Duration of CR were summarized using Kaplan-Meier estimates (median time, 95% CI for median time).
Time Frame: as for outcome 6
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox. Here, the "Overall Number of Participants Analyzed" denotes the number of participants who had achieved CR and had the first documented non-CR till end of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 9
months |  | NA [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | 25.89 [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | 70.34 [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). |  | 42.35 [17.45 to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed).

14. Primary Outcome: Duration of Objective Response
Description: Duration of response was measured from the first documentation of objective response (OR) to the first documented non-response of SD, PD, or relapse and was only evaluated in participants who had achieved an OR (CR or PR). Duration of OR was summarized using Kaplan-Meier estimates (median time, 95% CI for median time).
Time Frame: as for outcome 6
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox. Here, the "Overall Number of Participants Analyzed" denotes the number of participants who had achieved an OR (CR or PR) and had the first documented non-response of SD, PD, or relapse.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 6
months | 8.34 [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | 84.44 [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | 80.95 [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | 78.29 [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). |  | NA [52.11 to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed).

15. Primary Outcome: Time to Progression
Description: Time to disease progression/relapse is measured from the start of moxetumomab pasudotox treatment until the first documentation of disease progression or relapse and was summarized using Kaplan-Meier estimates (median time, 95% CI for median time).
Time Frame: as for outcome 6
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
months | 11.33 [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | NA [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | NA [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | 82.07 [2.00 to 82.07] | NA [0.92 to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | NA [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed).

16. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was measured from the start of moxetumomab pasudotox treatment until the first documentation of disease progression/relapse or death, whichever occurred first. PFS was summarized using Kaplan-Meier estimates (median time, 95% CI for median time).
Time Frame: as for outcome 6
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
months | 11.33 [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | NA [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | NA [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | 82.07 [2.00 to 82.07] | NA [0.92 to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed). | NA [NA to NA] — Not estimable because insufficient number of participants have events (progressed or relapsed).

17. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Moxetumomab Pasudotox for Cycle 1 on Day 1
Description: The Tmax is the time to reach maximum observed plasma concentration of Moxetumomab Pasudotox.
Time Frame: Cycle 1 Day 1: pre-infusion; at 15 minutes (min) during the infusion; at the end of infusion (approximately 5-7 minutes before the end of infusion); and at 1, 1.5, 2, 4, 8, and 12 hours (h) post infusion
Population: The PK Population consisted of all participants who received any amount of moxetumomab pasudotox and had a sufficient number of serum concentration measurements for computing PK parameters. The "Overall Number of Participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Median (Full Range); unit: hours
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 2 | 3 | 2 | 2 | 4 | 11
hours | 0.508 [0.383 to 0.633] | 0.467 [0.450 to 0.483] | 0.367 [0.233 to 0.500] | 0.467 [0.417 to 0.517] | 0.267 [0.250 to 0.417] | 0.417 [0.250 to 0.500]

18. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Moxetumomab Pasudotox for Cycle 1 on Day 5
Description: The Tmax is the time to reach maximum observed plasma concentration of Moxetumomab Pasudotox.
Time Frame: Cycle 1 Day 5: pre infusion; at 15 min during the infusion, at the end of infusion (approximately 5-7 minutes before the end of infusion); and at 1, 1.5, 2, 4, 8, and 12 h post infusion
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 4 | 12
hours | 0.500 [0.250 to 0.550] | 0.467 [0.417 to 0.483] | 0.250 [0.250 to 0.533] | 0.517 [0.417 to 0.617] | 0.475 [0.417 to 1.00] | 0.417 [0.283 to 0.517]

19. Primary Outcome: Maximum Observed Serum Concentration (Cmax) for Moxetumomab Pasudotox for Cycle 1 on Day 1
Description: The Cmax is the maximum observed plasma concentration of Moxetumomab Pasudotox.
Time Frame: Cycle 1 Day 1: pre-infusion; at 15 min during the infusion; at the end of infusion (approximately 5-7 minutes before the end of infusion); and at 1, 1.5, 2, 4, 8, and 12 h post infusion
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 4 | 12
nanogram per milliliter (ng/mL) | 77.5 (70.0) | 86.3 (41.9) | 49.4 (46.3) | 443 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 290 (107) | 435 (260)

20. Primary Outcome: Maximum Observed Serum Concentration (Cmax) for Moxetumomab Pasudotox for Cycle 1 on Day 5
Description: The Cmax is the maximum observed plasma concentration of Moxetumomab Pasudotox.
Time Frame: as for outcome 18
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 12
ng/mL | 103 (40.5) | 135 (49.1) | 161 (136) | 420 (384) | 701 (328) | 738 (316)

21. Primary Outcome: Area Under the Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC[0-last]) of Moxetumomab Pasudotox for Cycle 1 on Day 1
Description: The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Time Frame: as for outcome 19
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 2 | 3 | 2 | 2 | 4 | 11
nanogram*hour per milliliter (ng*h/mL) | 113 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 31.0 (20.9) | 109 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 897 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 183 (146) | 558 (590)

22. Primary Outcome: Area Under the Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC[0-last]) of Moxetumomab Pasudotox for Cycle 1 on Day 5
Description: The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Time Frame: as for outcome 18
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 4 | 12
ng*h/mL | 179 (155) | 90.2 (52.3) | 93.2 (113) | 1360 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 1640 (1270) | 1920 (1290)

23. Primary Outcome: Systemic Clearance (CL) of Moxetumomab Pasudotox for Cycle 1 on Day 1
Description: Systemic Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by area under plasma concentration-time curve from time zero to infinite time (AUC[0-infinity]).
Time Frame: as for outcome 19
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Milliliter/kilogram/hour (mL/kg/h)
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 2 | 0 | 1 | 2 | 1 | 8
Milliliter/kilogram/hour (mL/kg/h) | 32.6 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. |  | 49.1 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 43.9 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 91.8 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 106 (80.2)

24. Primary Outcome: Systemic Clearance (CL) of Moxetumomab Pasudotox for Cycle 1 on Day 5
Description: Systemic Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by AUC(0-infinity).
Time Frame: as for outcome 18
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mL/kg/h
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 4 | 10
mL/kg/h | 13.3 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 68.9 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 66.3 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 18.7 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 45.5 (47.6) | 33.3 (37.5)

25. Primary Outcome: Terminal Phase Elimination Half Life (t1/2) of Moxetumomab Pasudotox for Cycle 1 on Day 1
Description: The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Time Frame: as for outcome 19
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 2 | 0 | 1 | 2 | 1 | 8
hours | 0.643 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. |  | 3.77 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 1.00 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 0.375 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 0.799 (0.755)

26. Primary Outcome: Terminal Phase Elimination Half Life (t1/2) of Moxetumomab Pasudotox for Cycle 1 on Day 5
Description: as for outcome 25
Time Frame: as for outcome 18
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 4 | 10
hours | 2.20 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 0.369 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 0.404 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 1.86 (NA) — Standard deviation was reported only when the number of participants analyzed were >= 3. | 1.66 (0.928) | 2.06 (0.980)

27. Primary Outcome: AUC Accumulation Ratio of Moxetumomab Pasudotox for Cycle 1
Description: The AUC accumulation ratio of moxetumomab pasudotox was calculated as the geometric mean ratio of AUC(0-last) on the last day and the first day of a multiple dose regimen: Day 5/Day 1.
Time Frame: Cycle 1 Day 1 and Day 5: pre-infusion, at 15 min during the infusion, at the end of infusion, and at 1, 1.5, 2, 4, 8, and 12 h post infusion
Population: as for outcome 17
Measure: Median (Full Range); unit: ratio
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 2 | 3 | 2 | 2 | 4 | 11
ratio | 2.62 [1.22 to 4.02] | 3.08 [2.61 to 3.39] | 3.09 [0.0328 to 6.15] | 1.93 [1.20 to 2.66] | 12.4 [1.99 to 25.0] | 3.63 [1.73 to 21.8]

28. Primary Outcome: Cmax Accumulation Ratio of Moxetumomab Pasudotox for Cycle 1
Description: The Cmax accumulation ratio of moxetumomab pasudotox was calculated as the geometric mean ratio of Cmax on the last day and the first day of a multiple dose regimen: Day 5/Day 1.
Time Frame: as for outcome 27
Population: as for outcome 17
Measure: Median (Full Range); unit: ratio
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 2 | 3 | 2 | 2 | 4 | 11
ratio | 1.11 [0.934 to 1.29] | 1.73 [1.39 to 1.73] | 2.12 [0.839 to 3.40] | 1.48 [1.30 to 1.66] | 2.51 [1.47 to 3.26] | 1.58 [1.09 to 3.94]

29. Secondary Outcome: Number of Participants With Positive Neutralizing Antibodies and Correlation to Antitumor Activity
Description: Participants tested for immunogenicity to moxetumomab pasudotox prior to enrollment, before each cycle and at end of study. The neutralization assay measures the capacity of participant's plasma (antibodies) to inhibit the binding of moxetumomab pasudotox to its target, cluster of differentiation 22 (CD22), coated onto enzyme linked immunosorbent assay (ELISA) plates. Significant level of neutralizing antibody activity defined as the capacity of test plasma to inhibit >50% of the binding of CAT-8015 to CD22 using an ELISA-based method.
Time Frame: Up to end of treatment (approximately 8 years)
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
Participants | 2 | 2 | 2 | 1 | 0 | 7

30. Secondary Outcome: CD22 Expression Levels From Peripheral Blood by Best Response
Description: Participants malignant cells (peripheral blood) were tested for cluster of differentiation 22 (CD22) expression by fluorescence-activated cell sorter (FACS) analysis.
Time Frame: Prior to enrollment during screening, and for participants still having malignant cells, the test was to be repeated prior to each cycle of therapy, at the end of treatment, and end of the study (approximately 8 years)
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Mean (Standard Deviation); unit: sites per cell
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
sites per cell
  Peripheral Blood: Complete Response: number analyzed (Participants) | 0 | 1 | 2 | 1 | 1 | 18
  Peripheral Blood: Complete Response |  | 65434.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 72632.0 (12010.9) | 43803.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 61773.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 68141.3 (13614.0)
  Peripheral Blood: Partial Response: number analyzed (Participants) | 3 | 1 | 0 | 1 | 1 | 7
  Peripheral Blood: Partial Response | 38402.7 (14131.9) | 78356.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. |  | 76264.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 52495.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 33259.9 (25479.5)
  Peripheral Blood: Stable Disease: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 3
  Peripheral Blood: Stable Disease |  |  | 38939.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 84157.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. |  | 46089.3 (9644.6)
  Peripheral Blood: ProgressiveDisease: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Peripheral Blood: ProgressiveDisease |  |  |  |  | 24645.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. |

31. Secondary Outcome: CD22 Expression Levels From Bone Marrow by Best Response
Description: Participants malignant cells (paraffin block biopsy specimen) were tested for CD22 expression by FACS analysis.
Time Frame: as for outcome 30
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Mean (Standard Deviation); unit: sites per cell
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
sites per cell
  Bone Marrow: Complete Response: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 10
  Bone Marrow: Complete Response |  | 75157.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. |  | 50190.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. |  | 55850.5 (18482.2)
  Bone Marrow: Partial Response: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2
  Bone Marrow: Partial Response | 36286.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. |  |  |  |  | 37732.5 (9918.6)
  Bone Marrow: Stable Disease: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 2
  Bone Marrow: Stable Disease |  |  |  | 80400.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. |  | 36767.5 (720.5)
  Bone Marrow: Progressive Disease: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Soluble CD22 Levels by Best Response
Description: Soluble CD22 was collected from the participant's plasma and was performed at the NCI using an ELISA method.
Time Frame: as for outcome 30
Population: Safety population included all participants who received any treatment of moxetumomab pasudotox.
Measure: Mean (Standard Deviation); unit: picogram/mL
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 33
picogram/mL
  Complete Response: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 19
  Complete Response |  | 2583.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 60021.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 5109.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 10232.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 22202.9 (27809.4)
  Partial Response: number analyzed (Participants) | 3 | 1 | 0 | 1 | 3 | 6
  Partial Response | 3016.3 (1821.3) | 16675.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. |  | 5122.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 18238.5 (45.5) | 39493.5 (31216.9)
  Stable Disease: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0 | 4
  Stable Disease |  |  | 184750.0 (21566.8) | 528000.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. |  | 134129.5 (150498.4)
  Progressive Disease: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  Progressive Disease |  |  |  |  | 7484.0 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. |

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 30 days after the last dose of study drug (approximately 8 years)
Arm/Group | 5 mcg/kg | 10 mcg/kg | 20 mcg/kg | 30 mcg/kg | 40 mcg/kg | 50 mcg/kg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 2/3 | 0/4 | 4/33
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mcg/kg (N=3) | 10 mcg/kg (N=3) | 20 mcg/kg (N=3) | 30 mcg/kg (N=3) | 40 mcg/kg (N=4) | 50 mcg/kg (N=33)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mcg/kg (N=3) | 10 mcg/kg (N=3) | 20 mcg/kg (N=3) | 30 mcg/kg (N=3) | 40 mcg/kg (N=4) | 50 mcg/kg (N=33)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 25 (62)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 13 (21)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Chills (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 10 (17)
Fatigue (General disorders) | 1 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 8 (10)
Oedema (General disorders) | 1 (3) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 8 (10)
Oedema peripheral (General disorders) | 1 (5) | 1 (1) | 1 (1) | 3 (8) | 3 (7) | 13 (22)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (4) | 3 (5) | 1 (1) | 15 (25)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 7 (8)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (2) | 1 (3) | 3 (5) | 2 (5) | 25 (72)
Aspartate aminotransferase increased (Investigations) | 2 (7) | 1 (1) | 1 (3) | 2 (4) | 1 (4) | 24 (63)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (10)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Blood bilirubin increased (Investigations) | 2 (4) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 10 (19)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 2 (2)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (11)
Haemoglobin decreased (Investigations) | 2 (3) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 9 (15)
Haptoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (8)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 2 (7) | 5 (9)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (14)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (9)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
White blood cell count decreased (Investigations) | 2 (2) | 1 (1) | 2 (4) | 1 (3) | 2 (2) | 17 (23)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 13 (22)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 12 (20)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 19 (31)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (7) | 1 (1) | 1 (2) | 3 (9) | 3 (9) | 25 (72)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 11 (18)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 7 (15)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 3 (4) | 7 (10)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 10 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (3) | 0 (0) | 3 (7) | 2 (3) | 20 (36)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (10)
Headache (Nervous system disorders) | 1 (3) | 1 (1) | 1 (4) | 2 (3) | 1 (7) | 13 (21)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 8 (9)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 8 (10)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (8)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 10 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.